CLINICAL TRIAL: NCT07359586
Title: Incidence,Perioperative Risk Factors and Prognosis Associated With Laryngopharyngea Injury After Endotracheal Intubation Under General Anesthesia：A Retrospective Study
Brief Title: Laryngopharyngeal Injury After Endotracheal Intubation Under General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Other Study IDs: ZJU2025B0596
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Hepatic Carcinoma; Pulmonary Carcinoma; Pancreatic Carcinoma; Cholangiocarcinoma; Thyroid Carcinoma
Keywords: hoarseness; Vocal cord injury; Incidence; Prognosis
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Thyroid Neoplasms; Hoarseness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hoarseness: We collected perioperative clinical data from the cohort, analyzed the associated risk factors for the occurrence of relevant symptoms, and investigated the prognosis.

SUMMARY:
This study retrospectively analyzed patients who underwent tracheal intubation under general anesthesia at the First Affiliated Hospital of Zhejiang University School of Medicine between October 1, 2015, and September 30, 2025, with a focus on issues related to postoperativelaryngopharyngeal complaints. Patients requiring otolaryngological consultation due to postoperative laryngopharyngeal complaints were identified via the case consultation system. Relevant patient data were collected through the Medison Anesthesia Information Management System and electronic medical record system, and telephone follow-up was conducted to assess patient prognosis. The primary outcome measures were the risk factors of postoperative hoarseness, while the secondary outcome measures included the incidence of postoperative hoarseness, the severity of vocal fold injury and its related risk factors. Additionally, the prognosis of patients and its related risk factors were evaluated. This study aims to reduce the incidence of perioperative laryngopharyngeal injury and provide a reference for the optimization of perioperative anesthetic regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent general anesthesia with tracheal intubation at the First Affiliated Hospital of Zhejiang University School of Medicine between October 2015 and September 2025
* Patients who required otolaryngological consultation due to laryngopharyngeal complaints (including hoarseness, sore throat, cough, choking on drinking water, etc.) postoperatively
* The surgical type was non-otolaryngological surgery

Exclusion Criteria:

* Patients with a history of laryngopharyngeal lesions (e.g., granuloma, polyp, tumour, vocal cord paralysis
* Patients with a preexisting tracheotomy
* Patients requiring postoperative tracheotomy
* Patients with incomplete medical records
* Patients who underwent multiple surgeries but for whom the specific surgical episode responsible for the laryngopharyngeal complaints could not be identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent endotracheal intubation under general anesthesia at the First Affiliated Hospital of Zhejiang University between October 1, 2015, and September 30, 2025
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative hoarseness | Perioperative,up to150 days
  The patients underwent general anesthesia with tracheal intubation and required otolaryngological consultation for hoarseness between October 1, 2015, and September 30, 2025.Hoarseness is characterized by alterations in voice quality, pitch (how high or low the voice is), volume (loudness), or vocal effort that impair effective communication, as judged by a healthcare provider, and may adversely affect quality of life.

SECONDARY OUTCOMES:
Incidence of Hoarseness | Perioperative,up to150 days
  (Number of patients with postoperative hoarseness） / (Total number of patients undergoing general anesthesia tracheal intubation) × 100%
the severity of hoarseness | Perioperative,up to150 days
  Hoarseness was assessed as follows: 0 = none (no hoarseness), 1 = noticed by patient, 2 = obvious to observer, 3 = aphonia.
Postoperative Vocal Fold Injury | Perioperative,up to150 days
  Based on patients' hoarseness symptoms and laryngoscopic findings, an otolaryngologist conducted clinical assessment and grading, classifying vocal fold injury into four levels. The classification criteria were: Grade 0 (Normal): Non-hoarsenes; Grade 1 (Mild): hoarseness with negative laryngoscopic findings or vocal fold closure gap; Grade 2 (Moderate): hoarseness with vocal fold mobility impairment; Grade 3 (Severe): hoarseness with vocal cord paralysis or fixation.
Incidence of Arytenoid Dislocation | Perioperative,up to150 days
  (Number of patients with postoperative arytenoid dislocation)/ (Total number of patients undergoing general anesthesia tracheal intubation) × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - he First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided